CLINICAL TRIAL: NCT06123377
Title: Use of Angiogenic Factors in the Conservative Management of Gestational Hypertension. Prospective, Randomised, Controlled Study.
Brief Title: Angiogenic Factors in the Conservative Management of Gestational Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of the research deparment, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FA022023
Record Dates: First submitted 2023-10-29; First posted 2023-11-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Gestational Hypertension
Keywords: Gestational hypertension; Angiogenic factors
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 39 weeks (Experimental): Patients with gestational hypertension and angiogenic factors (sFlt-1/PIGF) below 33 will be evaluated weekly until 39 weeks, when termination of pregnancy will be scheduled.
  Interventions: Diagnostic Test: Angiogenic factor
- 37 weeks (Active Comparator): Patients with gestational hypertension and angiogenic factors (sFlt-1/PIGF) below 33 will be evaluated weekly until 37 weeks, when termination of pregnancy will be scheduled.
  Interventions: Diagnostic Test: Angiogenic factor

INTERVENTIONS:
Diagnostic Test: Angiogenic factor — sFLt-1/PGIF below or equal to 33

SUMMARY:
Hypertensive disorders of pregnancy (HPT) are an important cause of maternal-feto-neonatal morbidity and mortality, being one of the three leading causes of maternal death in our country and in developing countries. The only cure for THE is termination of pregnancy, which ends up being a decision in which gestational age and maternal risks must be balanced. Angiogenic factors have come to occupy an indispensable place in the arsenal of tools that can be used to separate the patient with a high likelihood of complications from those in whom prolongation of pregnancy could represent an important neonatal benefit. One of the most controversial scenarios is gestational hypertension, a group of hypertensive disorders considered the mildest form of the pre-eclamptic spectrum, where current recommendations indicate termination of pregnancy at 37 weeks. However, the decision is based on outdated guidelines developed at a time when angiogenic factors were just beginning to be known. The purpose of the study is to use angiogenic factors as a guide to decide the most appropriate gestational age for termination of pregnancy in patients diagnosed with gestational hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24 and 40 weeks of gestation.
* Diagnosis of Gestational Hypertension based on ACOG criteria
* index sFlt-1/PIGF equal or below 33

Exclusion Criteria:

* Multiple gestation
* Maternal vasculitis
* Previous cesarean section (3 or more)
* Neurological conditions
* Chronic renal disease
* Purpura
* Heart disease
* Index sFlt-1/PIGF of 34 or more

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression to preeclampsia | From the moment of randomization up until delivery. Between 1 and 17 weeks.
  In subject with gestational hypertension and sFlt-1/PIGF at enrollment equal or below 33, the appearance of proteinuria, severe criteria or sFlt-1/PIGF above 34

SECONDARY OUTCOMES:
Maternal / fetal morbidity | Up until discharge. On average, 7 days
  Presence of any/several indicators of maternal or fetal morbidity (abruptio placenta, HELLP syndrome, eclampsia, fetal growth restriction, acute lung edema).
Neonatal morbidity | Up until discharge. On average, 3 days
  Presence of any/several indicators of neonatal morbidity (Apgar scores, admission to NICU, encephalopatic hypoxia)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santo Tomas, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: Undecided